CLINICAL TRIAL: NCT03167450
Title: Examining the Knowledge, Attitudes, and Beliefs of Sickle Cell Disease Patients, Parents of Patients With Sickle Cell Disease, and Providers Towards the Integration of CRISPR in Clinical Care
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917081; 17-HG-N081
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Sickle Cell Disease
Keywords: CRISPR; Gene Editing; Qualitative; Participation Clinical Trials; Genetic Literacy
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Adults: Adults have sickle cell disease
- Parents: Parents with children/adults who have sickle cell disease
- Physicians: Physicians who have delivered healthcare to individuals living with sickle cell disease for at least a year

SUMMARY:
Background:

Sickle cell disease (SCD) is caused by a genetic defect that affects how hemoglobin is made. Due to this, people with SCD have abnormally-shaped red blood cells, which can result in poor oxygen transport in the body and increase risk of blood clots. CRISPR Cas9 is a new tool which allows scientists to snip and edit genes in a way that is faster, cheaper, and more precise than other gene-editing tools. Recently, research has been done using CRISPR Cas9 to correct the sickle cell gene in animal models and human cells. Researchers want to understand the views of those with SCD, parents of people with SCD, and the providers of these patients regarding use of CRISPR Cas9 in clinical trials and treatment.

Objectives:

To study the attitudes, beliefs, and opinions of those with SCD, parents of those with SCD, and providers on the use of CRISPR Cas9 gene-editing. An additional purpose of this study is to assess the utility of an educational tool for improving understanding of CRISPR Cas9.

Eligibility:

People ages 18 and older who speak English and either have SCD, are a parent of someone with SCD, or are a physician for people with SCD.

Design:

Participants will be screened via phone. Those with SCD will be screened with data from their SCD genotype.

Participation lasts about 2 hours.

Participants will fill out three surveys.

Participants will watch a video about CRISPR Cas9.

Participants will engage in a focus group session. This will be audiotaped and analyzed.

The data from the survey questions and focus groups may be used for future research. However, all personally identifiable information will be removed before data is shared.

Participants data will be identified with a code number instead of their name.

Participants may be invited to join future studies of SCD.

DETAILED DESCRIPTION:
The CRISPR/Cas9 gene-editing technique is taking the scientific research and healthcare community by storm with the promise it holds to cure and ease the burden of debilitating diseases. However, there is limited knowledge regarding the implications of using this type of tool in human research and medicine. Researchers need to understand the viewpoints of patients, their families, and their providers, to ensure that the approach taken towards gene-editing is inclusive and respectful of different interests and concerns. The dialogue, thus far, has been dominated by scientific researchers, physician scientists, ethicists, public health and policy experts. It is important to the advancement of the science to study the patient s perspective about the use of the technology. In addition, parents often play important roles in the decision-making process; in this regard, understanding the views and questions of this group of individuals regarding CRISPR/Cas9 human use is essential. We conduct a qualitative study with a mixed methods component to investigate the knowledge, attitudes and beliefs of patients living with sickle cell disease (SCD), the parents of patients with SCD, and the physicians of this patient population regarding the use of CRISPR/Cas9 technology. The study is designed to measure these three cohorts baseline overall genetic literacy, CRISPR-specific literacy, and general attitudes and beliefs toward gene-editing/CRISPR Cas9(in both somatic and germline cells); to evaluate the utility of an educational tool in improving one s understanding of this innovative technique; and to gauge how attitudes and beliefs toward gene-editing, specifically CRISPR Cas9, perhaps shift or remain intact after the educational video, as well as within a focus group space.

ELIGIBILITY:
* INCLUSION CRITERIA:

The inclusion criteria for patients:

1. must have a diagnosis of sickle cell disease
2. must be 18 years or older
3. must be English-speaking

The inclusion criteria for parents of patients with SCD:

1. must have a child with sickle cell disease
2. must be 18 years or older
3. must be English speaking

Lastly, the inclusion criteria for physicians:

1. must care for sickle cell patients
2. must have cared for sickle cell patients for a minimum of 12 months
3. must have been the caregiver for at least five adult patients and/or five pediatric patients
4. must be 18 years or older
5. must be English-speaking.

The participants need to be 18 years or older in order to provide informed consent. It is necessary that participants speak English due to the nature of the study. Because a moderated conversation will take place, it is essential that all participants and researchers speak the same language to allow for interactive discourse and comprehension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with sickle cell disease; parent of a child with sickle cell disease or physicians who have delivered healthcare to individuals living with sickle cell disease for at least a year
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Focus group interviews related to attitudes, beliefs, and opinions of those with SCD, parents of those with SCD, and providers on the use of CRISPR Cas9 gene-editing. | At the day of inclusion
To assess the utility of an educational tool for improving understanding of CRISPR Cas9. | At the day of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Vence L Bonham, J.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States